CLINICAL TRIAL: NCT01819597
Title: EDAS (Surgical) Revascularization for Symptomatic Intracranial Arterial Stenosis
Brief Title: Surgical Indirect Revascularization For Symptomatic Intracranial Arterial Stenosis
Acronym: ERSIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nestor R. Gonzalez, MD, MSCR., Professor of Neurosurgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23NS079477-01A1 (NIH)
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Intracranial Arterial Stenosis; Intracranial Atherosclerosis; Ischemic Stroke; Cerebral Angiogenesis
Keywords: Intracranial Arterial Stenosis; Atherosclerosis; Stroke; EDAS; Angiogenesis
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke; Atherosclerosis; Stroke

STUDY DESIGN:
Intervention Model Description: EDAS surgery for Intracranial atherosclerosis. Non-futility design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EDAS surgery (Other): EDAS surgery is an established form of indirect revascularization. The study arm in this study will receive EDAS surgery
  Interventions: Procedure: Encephaloduroarteriosynangiosis (EDAS)

INTERVENTIONS:
Procedure: Encephaloduroarteriosynangiosis (EDAS) — The operation is a form of indirect revascularization or EC-IC bypass, performed under general endotracheal anesthesia, with intraoperative electroencephalographic monitoring. The surgery consists in the dissection and relocation of the superficial temporal artery (STA) and middle meningeal artery (MMA) branches, which are separated from their surrounding tissues under microscopic visualization and re-routed through a craniotomy to be placed intracranially in close proximity to the branches of the middle cerebral artery (MCA). The MCA branches are dissected in the arachnoid space and the STA and MMA are kept in position with microsutures to the arachnoid or MMA dural cuffs, maintaining close contact between the EC and MCA branches.
  Other Names: Indirect revascularization; Indirect bypass; EC-IC revascularization; EC-IC indirect bypass; EC-IC indirect revascularization

SUMMARY:
Stroke due to intracranial arterial atherosclerosis is a significant medical problem, carrying one of the highest rates of recurrent stroke despite best medical therapy, with annual recurrence rates as elevated as 25% in high risk groups.

The goal of this investigation is to advance a promising surgical treatment for symptomatic atherosclerotic intracranial stenosis - encephaloduroarteriosynangiosis (EDAS). The investigation will test in a phase II futility trial the potential of EDAS for further development before proceeding with the design of a definitive clinical trial of EDAS Revascularization in patients with Symptomatic Intracranial Arterial Stenosis (ERSIAS).

The investigation is a 4-year futility trial to test the hypothesis that EDAS revascularization combined with aggressive medical therapy warrants further evaluation in a subsequent pivotal trial as an alternative to aggressive medical management alone for preventing the primary endpoint of stroke or death in patients with symptomatic intracranial arterial stenosis (Specific Aim 1). During the investigation the time course of collateralogenesis and perfusion improvement following EDAS will also be evaluated (Specific Aim 2.

DETAILED DESCRIPTION:
Intracranial arterial atherosclerosis is a significant medical problem, with elevated rates of recurrent stroke despite medical therapy, with annual recurrence rates for ischemic stroke reported in the SAMMPRIS Trial as high as 12.2% in the intensive medical therapy arm. The incidence of recurrence stroke can be even higher in some high-risk groups, as high as 25% in African-Americans and females. The ultimate goal of this project is to advance a promising surgical treatment for symptomatic atherosclerotic intracranial stenosis - encephaloduroarteriosynangiosis (EDAS). Compared with direct revascularization operations (bypass), EDAS has the advantages of being less technically demanding, avoiding temporary occlusion of cerebral vessels, and allowing gradual development of collateral circulation where the brain demands it, deterring early hyperperfusion and hemorrhage. There has been no systematic trial exploring the use of EDAS in cases of symptomatic, non-moyamoya intracranial arterial stenosis. Based on preliminary positive results, the investigators propose the long-term objective of demonstrating that EDAS improves the outcome in patients with symptomatic intracranial stenosis compared with aggressive medical therapy. This will require future phase III clinical trials. The present proposal has the purpose of testing in a phase II futility-design trial the potential of EDAS for further development before proceeding with the design of a definitive clinical trial of EDAS Revascularization in patients with Symptomatic Intracranial Arterial Stenosis (ERSIAS). The present project will be 4-year futility-design trial to determine if EDAS revascularization combined with aggressive medical therapy warrants further evaluation in a subsequent pivotal trial as an alternative to aggressive medical management alone for preventing the primary endpoint of stroke or death at two years in patients with symptomatic intracranial arterial stenosis (Specific Aim 1). During the investigation the investigators will systematically evaluate the time course of collateralogenesis and perfusion improvement following EDAS by using quantitative and semiquantitative perfusion MRI studies (Specific Aim 2). The new knowledge generated by this study on understanding the role of collateral circulation in stroke pathophysiology, patient selection, and use of non-invasive imaging will be useful not only for EDAS evaluation but potentially next generation stents and future novel medical therapies, such as use of angiogenic growth factors and/or endothelial stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. TIA or non-severe stroke within 30 days of enrollment attributed to 70% to 99% stenosis* of a major intracranial artery (carotid artery or MCA)

   *May be diagnosed by TCD, MRA, or CTA to qualify, but must be confirmed by catheter angiography as per usual clinical practice.
2. Modified Rankin scale score of ≤3
3. Target area of stenosis in an intracranial artery that has a normal diameter of 2.00 mm to 4.50 mm
4. Target area of stenosis is ≤14 mm in length
5. Age ≥30 years and ≤80 years

   * Patients 30 to 49 years of age are required to meet at least 1 additional criteria (i-vi) provided below to qualify for the study. This additional requirement is to increase the likelihood that the symptomatic intracranial stenosis in patients 30 to 49 years is atherosclerotic: i. Insulin-dependent diabetes for at least 15 years ii. At least 2 of the following atherosclerotic risk factors: hypertension (BP ≥ 140/90 mm Hg or on antihypertensive therapy); dyslipidemia (LDL ≥130 mg/dL or HDL ≤40 mg/dL or fasting triglycerides ≥150 mg/dL or on lipid lowering therapy); smoking; non-insulin-dependent diabetes or insulin-dependent diabetes of <15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, and peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event.

   iii. History of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease iv. Any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by noninvasive vascular imaging or catheter angiography and is considered atherosclerotic v. Aortic arch atheroma documented by noninvasive vascular imaging or catheter angiography vi. Any aortic aneurysm documented by noninvasive vascular imaging or catheter angiography that is considered atherosclerotic
6. Negative pregnancy test in a female who has had any menses in the last 18 months
7. Patient is willing and able to return for all follow-up visits required by the protocol.
8. Patient is available by phone.
9. Patient understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent.
10. Demonstration of poor or no collateral flow in the territory of the qualifying stenotic vessel (ASITN/SIR Collateral Flow Grades 0-2) and hypoperfusion of the vascular territory in MRI.

Exclusion Criteria:

1. Tandem extracranial or intracranial stenosis (70-99%) or occlusion that is proximal or distal to the target intracranial lesion
2. Bilateral intracranial vertebral artery stenosis of 70% to 99% and uncertainty about which artery is symptomatic (e.g., if patient has pontine, midbrain, or temporal occipital symptoms)
3. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days before the expected enrollment date
4. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform staged angioplasty followed by stenting of target lesion
5. Plan to perform concomitant angioplasty or stenting of an extracranial vessel tandem to an intracranial stenosis
6. Presence of intraluminal thrombus proximal to or at the target lesion
7. Any aneurysm proximal to or distal to the stenotic intracranial artery
8. Intracranial tumor (including meningioma) or any intracranial vascular malformation
9. Computed tomographic or angiographic evidence of severe calcification at target lesion
10. Thrombolytic therapy within 24 hours before enrollment
11. Progressive neurologic signs within 24 hours before enrollment
12. Brain infarct within previous 30 days of enrollment that is of sufficient size (> 5 cm) to be at risk of hemorrhagic conversion during or after surgery
13. Any hemorrhagic infarct within 14 days before enrollment
14. Any hemorrhagic infarct within 15 to 30 days that is associated with mass effect
15. Any history of a primary intracerebral (parenchymal) hemorrhage
16. Any other intracranial hemorrhage (subarachnoid, subdural, or epidural) within 30 days
17. Any untreated chronic subdural hematoma >5 mm in thickness
18. Intracranial arterial stenosis related to arterial dissection, Moya-Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid pleocytosis; radiation-induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process, and suspected recanalized embolus
19. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction <30%
20. Known allergy or contraindication to aspirin and local or general anesthesia
21. History of life-threatening allergy to contrast dye. If not life-threatening and can be effectively pretreated, patient can be enrolled at physician's discretion
22. Known absolute contraindication to obtaining MRI studies, such as magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neuro-stimulators, and cochlear implants), MRI incompatible orthopedic implants, and free metallic fragments in the brain or eye.
23. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets <100,000, hematocrit <30, INR >1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic BP>180 mm Hg or diastolic BP>115 mm Hg), severe liver impairment (AST or ALT > 3 times normal, cirrhosis), creatinine > 3.0 (unless on dialysis)
24. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 90 days after enrollment
25. Indication for warfarin or heparin beyond enrollment (NOTE: Exceptions allowed for use of subcutaneous heparin for deep venous thrombosis prophylaxis while hospitalized)
26. Severe neurologic deficit that renders the patient incapable of living independently
27. Dementia or psychiatric problem that prevents the patient from following an outpatient program reliably
28. Comorbid conditions that may limit survival to < 3 years
29. Females who are pregnant or of childbearing potential and unwilling to use contraception for the duration of this study
30. Enrollment in another study that would conflict with the current study

Surgical Specific Exclusion Criteria:

In addition to those enumerated above, given the surgical nature of the intervention for patients failing best medical therapy, the following are additional exclusion criteria:

1. Use of clopidogrel or extended release dipyridamole within 7 days of the date of surgery. This exclusion is based on the elevated risk of hemorrhagic complications for intracranial surgery using those agents according to the current AHA/ACC Guidelines (Fleisher et al., 2007).
2. Evidence of active, un-treated focal or systemic infections (i.e. pneumonia, urinary tract infection, skin abscess) or history of recurrent infections despite treatment in the last 6 months.
3. Coagulation disorders characterized by a PTT ≥ 34, or a PT ≥ 12, or an INR ≥ 1.3, or a platelet count of <80,000.
4. Non-controlled hyperglycemia (any pre-prandial glucose level ≥ 180 mg/dL in any single test within 30 days before enrollment) or a hemoglobin A1c (HbA1c) ≥7%.
5. A low-density lipoprotein cholesterol (LDL-c) ≥ 130 mg/dL.
6. A non-high-density lipoprotein cholesterol (non-HDL-c) ≥ 100 mg/dL.
7. Smoking history in the last 6 months.
8. BMI ≥ 30 kg/m2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor R Gonzalez, MD, MSCR, Principal Investigator — Cedars Sinai Neurosurgery
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Dusick JR, Liebeskind DS, Saver JL, Martin NA, Gonzalez NR. Indirect revascularization for nonmoyamoya intracranial arterial stenoses: clinical and angiographic outcomes. J Neurosurg. 2012 Jul;117(1):94-102. doi: 10.3171/2012.4.JNS111103. Epub 2012 May 4. PMID 22559848
- [Background] Gonzalez NR, Liebeskind DS, Dusick JR, Mayor F, Saver J. Intracranial arterial stenoses: current viewpoints, novel approaches, and surgical perspectives. Neurosurg Rev. 2013 Apr;36(2):175-84; discussion 184-5. doi: 10.1007/s10143-012-0432-z. Epub 2012 Oct 25. PMID 23097149
- [Background] Dusick JR, Gonzalez NR, Martin NA. Clinical and angiographic outcomes from indirect revascularization surgery for Moyamoya disease in adults and children: a review of 63 procedures. Neurosurgery. 2011 Jan;68(1):34-43; discussion 43. doi: 10.1227/NEU.0b013e3181fc5ec2. PMID 21150753
- [Derived] Gonzalez NR, Jiang H, Lyden P, Song S, Schlick K, Dumitrascu O, Quintero-Consuegra MD, Toscano JF, Liebeskind DS, Restrepo L, Rao N, Hinman J, Alexander MJ, Schievink W, Piantadosi S, Saver JL. Encephaloduroarteriosynangiosis (EDAS) revascularization for symptomatic intracranial atherosclerotic steno-occlusive (ERSIAS) Phase-II objective performance criterion trial. Int J Stroke. 2021 Aug;16(6):701-709. doi: 10.1177/1747493020967256. Epub 2020 Oct 29. PMID 33115382
- [Derived] Laiwalla AN, Ooi YC, Van De Wiele B, Ziv K, Brown A, Liou R, Saver JL, Gonzalez NR. Rigorous anaesthesia management protocol for patients with intracranial arterial stenosis: a prospective controlled-cohort study. BMJ Open. 2016 Jan 19;6(1):e009727. doi: 10.1136/bmjopen-2015-009727. PMID 26787251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at UCLA Medical Center and Cedars Sinai Medical Center in Los Angeles.
Groups:
- EDAS Surgery: EDAS surgery is an established form of indirect revascularization. The study arm in this study received EDAS surgery
  Encephaloduroarteriosynangiosis (EDAS): The operation is a form of indirect revascularization or EC-IC bypass, performed under general endotracheal anesthesia, with intraoperative electroencephalographic monitoring. The surgery consists in the dissection and relocation of the superficial temporal artery (STA) and middle meningeal artery (MMA) branches, which are separated from their surrounding tissues under microscopic visualization and re-routed through a craniotomy to be placed intracranially in close proximity to the branches of the middle cerebral artery (MCA). The MCA branches are dissected in the arachnoid space and the STA and MMA are kept in position with microsutures to the arachnoid or MMA dural cuffs, maintaining close contact between the EC and MCA branches.
Period: Overall Study
Arm/Group | EDAS Surgery
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Stroke or Death in the Territory of Qualifying Artery
Description: The primary study endpoint is the number of participants with any stroke or death within 30 days after enrollment, or any ischemic stroke or death attributable to ischemia in the territory of the qualifying artery at one year.
  Ischemic stroke is defined as a new focal neurological deficit of sudden onset, lasting at least 24 hours and not associated with CT or MRI findings of hemorrhage.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 5
Statistical Analysis 1: Comparison: EDAS Surgery; We derived the sample size required to power the trial to test the difference between two binomial event rates using the method of Farrington and Manning as implemented in R package gsDesign (Anderson, 2011). An estimated sample size of 52 patients will be necessary to detect a ∆ of 0.05, with a one-sided alpha of 0.10 and a beta of 0.10 - acceptable parameters for a non-definitive, non-futility study (Palesch et al., 2005, Levin, 2005); Test type: Other — This is a phase II study design to determine the non-futility of proceeding to a phase III pivotal evaluation. The study group was planned to be compared to a propensity score matching (PSM) cohort from to the patients in the medical arms of the SAMMPRIS trial and to patients in the medical arm of COSS that had demonstrated angiographic intracranial atherosclerosis and occlusion; p = 0.08, Regression, Cox — Pre-established α ≤ 0.10 for phase IIa; Alpha set at ≤ 0.1. for phase II study; Hazard Ratio (HR) = 0.38, 90% CI 2-sided [0.14 to 0.94] — ERSIAS/ Controls

2. Secondary Outcome: Myocardial Infarction
Description: Number of participants with heart attack within 30 days of surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 1

3. Secondary Outcome: Major Non-stroke Hemorrhage
Description: Number of participants with systemic hemorrhage, subdural or epidural hemorrhages
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 0

4. Secondary Outcome: Functional Outcome
Description: Proportion of participants with good functional outcome at the end of follow-up measured by the modified Rankin scale (mRS). That is with mRS scores between 0 and 2.
  Modified Rankin Scale
  Score and Description:
  0 - No symptoms at all
  1. - No significant disability despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. - Dead
Time Frame: 2 years
Population: Good functional outcome (Modified Rankin Scores 0-2)
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 45

5. Secondary Outcome: Cognitive Outcome
Description: Mean cognitive outcome at the end of follow-up measured by the Montreal Cognitive Assessment (MoCA). Scores on the MoCA scale range between 0 and 30. Higher values represent a better outcome. A normal score on the MoCA scale is 26 or higher.
Time Frame: 2 years
Population: Montreal Cognitive Outcome Assessment (MoCA)
Measure: Mean (Standard Deviation); unit: MoCA Score
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
MoCA Score | 25.5 (4.1)

6. Secondary Outcome: Improved Collaterals
Description: Number of participants with an increase by at least one grade on the American Society of Interventional and Therapeutic Neuroradiology/Society of Interventional Radiology (ASITN/SIR) Collateral Flow Grading System
  The ASITN/SIR Collateral Flow Grading System has 4 grades:
  0=no collaterals visible to the ischemic site.
  1. slow collaterals to the periphery of the ischemic site with persistence of some of the defect
  2. rapid collaterals to periphery of ischemic site with persistence of some of the defect and to only a portion of the ischemic territory
  3. collaterals with slow but complete angiographic blood flow of the ischemic bed by the late venous phase
  4. complete and rapid collateral blood flow to the vascular bed in the entire ischemic territory by retrograde perfusion.
  Grade 4 represents the best outcome. Grade 0 represents the worst outcome.
Time Frame: 1 year
Population: Evidence of angiographic neovasculariozation
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 41

7. Secondary Outcome: Asymptomatic Cerebral Hemorrhage
Description: Asymptomatic cerebral hemorrhage, defined as parenchymal or intraventricular bleeding detected in any imaging modality that is not associated with neurological deficits.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | EDAS Surgery
Number analyzed (Participants) | 52
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: All adverse events were adjudicated by independent neurologists not involved in the surgical procedure
Arm/Group | EDAS Surgery
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 2/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDAS Surgery (N=52)
Death with 30 days of surgery (Cardiac disorders) | 1 (1) — Death 28 days after the EDAS surgery in a 70 y/o patient who suffered a large myocardial infarction three weeks after surgery and secondary cardiac tamponade.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDAS Surgery (N=52)
Wound dehiscenece (Musculoskeletal and connective tissue disorders) | 2 (2) — Surgical wound dehiscence that required an additional surgical intervention for debridement and closure.

LIMITATIONS AND CAVEATS:
None. Trial was completed as planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT01819597/Prot_SAP_000.pdf